CLINICAL TRIAL: NCT03263533
Title: HDAC Inhibitor Augmentation to Clozapine
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PIs were unable to recruit any participants
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20007977
Record Dates: First submitted 2017-08-14; First posted 2017-08-28 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Schizophrenia
Keywords: schizophrenia; clozapine; vorinostat; HDAC; histone deacetylase inhibitor
MeSH Terms: conditions — Schizophrenia | interventions — Vorinostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vorinostat Group 1 (P-V-P-P) (Experimental): This group will receive this sequence after the 1 initial week washout:
  vorinstat (4 weeks) placebo (1 week) placebo (4 weeks)
  Interventions: Drug: Vorinostat Oral Capsule Group 1
- Vorinostat Group 2 (P-P-P-V) (Experimental): This group will receive this sequence after the 1 initial week washout:
  placebo (4 weeks) placebo (1 week) vorinostat (4 weeks)
  Interventions: Drug: Vorinostat Oral Capsule Group 2

INTERVENTIONS:
Drug: Vorinostat Oral Capsule Group 1 — Following the initial washout and first 4-week period of the trial, all patients will enter a second 1-week washout. After the washout, all patients will then enter a second 4 week alternate treatment (vorinostat or placebo). During the vorinostat sequence, doses will be increased over the first 2 weeks in each phase of the crossover study, starting by 100 mg per day, and increasing to 200 mg by week 2 and 300 mg per day at the start of week 3 until the end of week 4.
  Arms: Vorinostat Group 1 (P-V-P-P)
Drug: Vorinostat Oral Capsule Group 2 — Following the initial washout and first 4-week period of the trial, all patients will enter a second 1-week washout. After the washout, all patients will then enter a second 4 week alternate treatment (vorinostat or placebo). During the vorinostat sequence, doses will be increased over the first 2 weeks in each phase of the crossover study, starting by 100 mg per day, and increasing to 200 mg by week 2 and 300 mg per day at the start of week 3 until the end of week 4.
  Arms: Vorinostat Group 2 (P-P-P-V)

SUMMARY:
The main goal of this pilot study is to test the extent to which adjunctive treatment with the histone deacetylase (HDAC) inhibitor vorinostat improves brain plasticity and cognition in a pilot placebo-controlled trial in patients with schizophrenia who are on clozapine.

DETAILED DESCRIPTION:
The goal of this study is to perform a pilot clinical study with a small sample of subjects to evaluate the safety and tolerability of vorinostat when combined with clozapine treatment in patients with schizophrenia. The investigators will also evaluate the potential translation of our preclinical data into a clinical use of vorinostat for cognitive impairment in clozapine-treated schizophrenic patients.

Potential participants will be receiving stables doses of clozapine for a minimum period of 6 months before entry into the study. Clozapine was selected because i) the majority of our studies in mouse models were performed after chronic treatment with this atypical antipsychotic, and ii) the investigators' data in postmortem human brain samples of subjects with antemortem diagnosis of schizophrenia suggest up-regulation of HDAC2 in frontal cortex of schizophrenic subjects treated with atypical, but not typical, antipsychotic drugs.

The HDAC inhibitor vorinostat was selected because preliminary data suggest that chronic treatment with vorinostat improves HDAC2-dependent cognitive function in rodent models. Additionally, vorinostat is the first HDAC inhibitor approved by the U.S. Food and Drug Administration (FDA) for the treatment of cutaneous T-cell lymphoma. Dose(s) of vorinostat have been selected based on previous clinical studies in such patients with brain metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with DSM-5 Schizophrenia
* Receiving stable dose pf clozapine (≥ 300 mg per day) for at least 6 months before entering the study

Exclusion Criteria:

* Taking specific psychotropic medications (lamotrigine and valproic acid)
* Current or recent (12-months) substance use or induced disorder
* History of significant neurological or medical disorders
* Intellectual disability
* Known contraindications to the administration of vorinostat per product labeling
* Women currently pregnant, planning to become pregnant, or receiving hormone therapy and refusing any form of birth control

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 10 weeks
  Safety of vorinostat measured by number of adverse events
Change in clinical cognitive symptoms during adjunctive vorinostat therapy in schizophrenia patients treated with clozapine | Baseline, Visit 4 (end of first intervention group/week 4), Visit 7 (end of study/10 weeks)
  Participants will be given a cognitive test to assess executive function and speed.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Gonzalez-Maeso, PhD, Principal Investigator — Virginia Commonwealth University

IPD SHARING:
Plan to Share IPD: No